CLINICAL TRIAL: NCT03507816
Title: Epidemiology and Treatment of Multidrug-resistant (MDR TB) and Extensively Drug- Resistant (XDR TB) Tuberculosis in Strasbourg, France; a 10 Years Retrospective Study
Brief Title: A Multidrug-resistant (MDR) and Extensively Drug- Resistant (XDR) Tuberculosis Study in Alsace
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7002
Record Dates: First submitted 2018-02-16; First posted 2018-04-25 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Multi-drug Resistant Tuberculosis; Observational retrospective study; Clinical epidemiology; Treatment outcome; Migrant; Precarity
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine the epidemiology of TB MR in Strasbourg and evaluate the second-line anti-tuberculosis treatments effectiveness, and the relevance and adequacy of the treatments with WHO recommendations. During years 2006-2016, all new cases of MDR TB or XDR TB diagnosed Strasbourg University Hospital will be included in the study (22 cases). Data were collected from the Center for Tuberculosis Control (CLAT) records, the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years old)
* Patient hospitalized at Strasbourg University Hospital from 2006 to 2016, with proven MDR or XDR tuberculosis

Exclusion Criteria:

- Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with proven MDR or XDR tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Study of clinical characteristics of patients hospitalized at Strasbourg University Hospital from 2006 to 2016, with proven MDR or XDR tuberculosis | The period from January 1st, 2006 to December 31st, 2016 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ARGEMI, MD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Maladies Infectieuses et Tropicales, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No